CLINICAL TRIAL: NCT06961058
Title: In Person vs Telehealth Opioid Use Disorder Treatment After Patients Leave the Emergency Department
Brief Title: Telehealth vs In-Person Evaluation of Addiction Treatment After Visiting the Emergency Department
Acronym: TREATED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2262435; BPS-2023C3-35503 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
Keywords: emergency department; buprenorphine; telehealth; comparative effectiveness
MeSH Terms: conditions — Opioid-Related Disorders; Emergencies

STUDY DESIGN:
Intervention Model Description: Our study will use a two-stage randomization procedure. Patients will first be randomized 3:1 to either a "random assignment" group, which will then be further randomized 1:1 to one of the two arms, or a "patient choice" group. Patients in the "patient choice" group will be assigned to their preferred arm. If patients in this group have no preference, we will randomize them 1:1 to one of the arms. This approach allows estimation of both treatment effects and effects of patient preference on outcomes.
Masking Description: Research staff will be unaware of participant arm assignment until after the participant has enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- in person (Active Comparator): Participants will get treatment via CA Bridge, California's statewide program to provide Emergency Department (ED)-based OUD treatment. When clinicians or staff suspect an ED patient may have OUD, they refer the patient to an ED-based counselor who assesses the patient and engages them in OUD care. All patients with OUD get brief counseling and take-home naloxone. Patients willing to start treatment get buprenorphine (via either ED- or home-based induction), a referral for in-person outpatient OUD treatment at a local outpatient clinic or opioid treatment program, and a "bridge" prescription of buprenorphine to last until their first outpatient appointment. CA Bridge counselors maintain contact with patients for up to 30 days to help them establish outpatient care. This is usual care in study hospitals and in the >80% of California hospitals that participate in CA Bridge.
  Interventions: Other: referral to in person treatment
- telehealth (Experimental): This arm will comprise the same elements as the "in person" arm except that patients will be referred to get outpatient OUD treatment via telehealth (i.e. phone or video visits). Depending on study site and patient insurance, participants will be referred to get treatment at either a clinic associated with their hospital that offers telehealth OUD treatment or from a digital health company that provides on-demand telehealth OUD treatment and support services via video and phone visits.
  Interventions: Other: referral to telehealth treatment

INTERVENTIONS:
Other: referral to telehealth treatment — the intervention tested will be referral to get outpatient treatment via telehealth. Participants in the telehealth arm will receive the intervention.
  Arms: telehealth
Other: referral to in person treatment — participants in the in person arm will be referred to in person OUD treatment after they leave the ED
  Arms: in person

SUMMARY:
Main study objective: compare long-term buprenorphine treatment outcomes for patients who start buprenorphine for opioid use disorder (OUD) in the emergency department and are then referred to get outpatient buprenorphine treatment either via telehealth or at an in-person clinic.

Researchers will:

Compare rates of establishing outpatient OUD treatment, how long patients stay on buprenorphine, and patients' experience with care to determine whether patient experiences and outcomes are better for patients referred to telehealth treatment versus patients patients referred to in-person treatment after they leave the emergency department.

Participants will:

Be recruited from 3 different hospital emergency departments.

Answer questionnaires at baseline and then 1, 3, 6, and 9 months after their initial emergency department visit.

DETAILED DESCRIPTION:
Buprenorphine is a lifesaving but underused medication for treating opioid use disorder (OUD). Providing buprenorphine for OUD in hospital emergency departments is an evidence-based practice that reduces patients' risk of overdose. Most people with OUD need to stay on buprenorphine for years, yet median buprenorphine adherence is typically less than six months. There is thus a clear need for strategies to increase long term buprenorphine retention, particularly among patients prescribed buprenorphine in emergency departments, who often face barriers when transitioning to outpatient OUD treatment after they leave the emergency department. The practice of providing outpatient OUD treatment via telehealth (e.g., through video or phone visits) was developed years ago to serve rural areas, but it has become much more widely used and accepted across the US since the COVID-19 pandemic. Telehealth OUD treatment may also reduce logistical barriers to treatment (e.g., transportation) and reduce impacts of patient-reported OUD stigma (by reducing in-person visits to addiction clinics). This proposed study will address the following research question: For patients prescribed buprenorphine for OUD in hospital emergency departments and then referred for outpatient buprenorphine treatment, how do rates of establishing outpatient treatment and long-term retention in treatment compare for patients referred to treatment in person (at outpatient clinics or opioid treatment programs) versus treatment via telehealth? The study hypothesis is that rates of engaging with outpatient treatment, long-term buprenorphine retention, and patients' experience with care will be greater for patients referred to telehealth compared to in-person OUD treatment. To test this hypothesis, this project will conduct a pragmatic clinical trial at three emergency departments that participate in "CA Bridge," a statewide California program to encourage substance use treatment in emergency departments. Patients started on buprenorphine for OUD in the emergency department will be recruited and randomized 3:1 to either a random assignment group or a group where patients can choose their outpatient arm assignment. Patients in the random assignment group will be further randomized 1:1 to be referred to either in-person or telehealth outpatient treatment. This 2-step study design allows researchers to estimate both traditional effect sizes and the impact of patient preference on outcomes. Buprenorphine prescribing will be measured using prescription records from California's prescription drug monitoring program; patient questionnaires will be administered at baseline and 1, 3, 6, and 9 months after patients' emergency department visit. Treatment outcomes will be the proportion of patients establishing outpatient OUD treatment (i.e., filling at least one outpatient buprenorphine prescription within 30 days of their emergency department) and cumulative days with an active buprenorphine prescription six months after their emergency department visit (primary outcome). Drug related fatal overdose will be measured using California death certificate data. Subsequent emergency department visits and hospitalizations will be assessed from electronic health records. Patients' experience with care will be measured using AHRQ's Consumer Assessment of Health Providers and Systems Clinician and Group survey version 4.0, which includes questions specific to telehealth encounters. Finally, this study will examine associations between patients' baseline reports of OUD stigma and subsequent treatment outcomes as well as how arm assignment effects this association. Study findings will fill key evidence gaps and directly inform decisions by clinicians and patients about where patients should be referred for outpatient buprenorphine treatment after they leave the emergency department. Compared to the general population with OUD, patients who seek OUD care in the emergency department have higher overdose risk and are disproportionately low-income, non-white, and unstably housed. Thus, improving buprenorphine retention among patients who start treatment in the emergency department also has potential to reduce socioeconomic disparities in OUD treatment and, ultimately, overdose rates. Findings from our study will be immediately applicable to clinicians and patients in the nearly 300 hospital emergency departments across California that participate in the CA Bridge program as well as to hospitals across the country that have implemented emergency department-based OUD treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who present to the emergency department and receive buprenorphine (either administered or prescribed) to treat OUD
* do not have an established outpatient clinic where they will get buprenorphine when they leave the emergency department

Exclusion Criteria:

* inability to give consent
* patients living in institutions (e.g., nursing homes, prisons)
* unable to complete questionnaires in either English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
buprenorphine retention | 6 months
  cumulative days with an active buprenorphine prescription

SECONDARY OUTCOMES:
buprenorphine retention | 3 months, 9 months
  cumulative days with an active buprenorphine prescription
buprenorphine retention (binary) | 3, 6, 9 months
  active buprenorphine prescription with no gap in coverage >7 days
drug overdose death | 1, 3, 6, 9 months
  death related to overdose
past 30-day opioid use | 1, 3, 6, 9 months
  patient-reported number of days patient used opioids (illicit opioids or prescription opioids for non-medical reasons) during past 30 days
patient experience with care | 1, 3, 6, 9 months
  Access and visit rating subscales of AHRQ CAHPS clinician and group survey
non-fatal overdose | 1, 3, 6, 9 months
  non-fatal overdose related to drug use, assessed from a combination of patient report and hospital electronic health records
establishing outpatient treatment | 1 month
  patients filling at least 1 outpatient buprenorphine prescription within 30 days of their emergency department visit

OTHER OUTCOMES:
health care utilization | 1, 3, 6, 9 months
  emergency department visits and/or hospital admissions

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Moulin, MD MAS, Principal Investigator — University of California, Davis; Stephen G Henry, MD MSc, Principal Investigator — University of California, Davis
Locations (3):
- United States (3):
  - El Centro Regional Medical Center Emergency Department, El Centro, California
  - University of California Davis Emergency Department, Sacramento, California
  - Olive View - UCLA Medical Center Emegency Department, Sylmar, California

IPD SHARING:
Plan to Share IPD: No
sharing is not required by the study funder for this project

REFERENCES:
- [Background] D'Onofrio G, Chawarski MC, O'Connor PG, Pantalon MV, Busch SH, Owens PH, Hawk K, Bernstein SL, Fiellin DA. Emergency Department-Initiated Buprenorphine for Opioid Dependence with Continuation in Primary Care: Outcomes During and After Intervention. J Gen Intern Med. 2017 Jun;32(6):660-666. doi: 10.1007/s11606-017-3993-2. Epub 2017 Feb 13. PMID 28194688
- See also: PCORI (funder) website for this study — https://www.pcori.org/research-results/2024/person-versus-telehealth-opioid-use-disorder-treatment-after-patients-leave-emergency-department